CLINICAL TRIAL: NCT03751670
Title: Pulmonary Rehabilitation During Acute Exacerbations of Chronic Obstructive
Brief Title: Pulmonary Rehabilitation During Acute Exacerbations of Chronic Obstructive Pulmonary Disease: a Mixed-methods Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFRH/BD/147200/2019
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; Pulmonary rehabilitation; Community; Home
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR+conventional treatment (Experimental): Patients will be treated with daily medication prescribed by the physician. Additionally, patients will receive 6 sessions (2 times a week during 3 weeks) of Pulmonary Rehabilitation (PR). PR will include breathing retraining and airway clearance techniques, exercises for thoracic mobility, expansion and flexibility, cardiorespiratory exercise training, education and psychosocial support.
  Interventions: Other: Pulmonary Rehabilitation; Drug: Daily medical treatment
- Conventional treatment (Active Comparator): Patients will be treated with daily medication prescribed by the physician.
  Interventions: Drug: Daily medical treatment

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation programmes will include breathing retraining and airway clearance techniques, exercises for thoracic mobility, muscle strength, cardiorespiratory exercise training, education and psychosocial support.
  Arms: PR+conventional treatment
Drug: Daily medical treatment — Patients will be treated with daily medication prescribed by the physician.
  Other Names: Medication

SUMMARY:
This study aims to i) assess the short-, mid- and long-term effectiveness of a patient-centred community-based pulmonary rehabilitation (PR) programme during during acute exacerbations of chronic obstructive pulmonary disease (AECOPD); ii) establish the minimal clinical important differences for PR in AECOPD for clinical and patient-reported outcome measures; and iii) evaluate patients' perspectives and self-reported impact of the PR programme.

Patients with AECOPD will be recruited via clinicians at hospitals and primary care centres. Sociodemographic, anthropometric and clinical data; vital signs and peripheral oxygen saturation; symptoms (dyspnoea, fatigue, cough and sputum); lung function; physical activity level; peripheral muscle strength; functional status; exercise tolerance; impact of the disease and health-related quality of life will be collected within 24h-48h of the AECOPD diagnosis. Then, patients will be randomly allocated to either conventional treatment or conventional treatment plus PR. After 3 weeks, all outcome measures will be reassessed. Additionally, follow-ups at 2, 6 and 12 months will be performed through phone calls to assess the number of recurrent AECOPD, healthcare utilization and mortality.

Conventional treatment will consist on daily medical treatment prescribed by the physician (i.e., medication).

Community-based PR will involve 6 sessions (2 times per week) of breathing retraining and airway clearance techniques, exercises for thoracic mobility, expansion and flexibility, cardiorespiratory exercise training, education and psychosocial support.

It is expected that, by including PR in the treatment of patients with AECOPD, they will express greater improvements in a shorter period of time and experience a decrease number of re-exacerbations and healthcare utilization.

DETAILED DESCRIPTION:
Acute exacerbations of COPD (AECOPD) negatively impact on patients' health status and disease progression, and increase patients' susceptibility to exacerbations, hospitalizations and death. Therefore, the treatment goals for patients with AECOPD are to minimize the negative impact of these events and prevent their recurrence.

Pulmonary rehabilitation (PR) is the comprehensive intervention presenting the most well-established benefits in patients with stable COPD, thus, it would seem reasonable to consider PR as a management strategy for AECOPD. However, studies assessing PR role during AECOPD have shown conflicting results.

Therefore, the main aim of this project is to assess the short-, mid- and long-term effectiveness of a patient-centered community-based PR programme during AECOPD. Secondarily, we aim to develop and implement a community-based PR programme for patients with AECOPD, specifically tailored to their self-reported and clinical needs; establish the minimal clinical important differences for PR in AECOPD for clinical and patient-reported outcome measures; and evaluate patients' perspectives and self-reported impact of the PR programme.

A pilot study was performed between November 2016 and December 2017 to allow sample size calculation and adjustments to the protocol of the randomized controlled trial. Based on this pilot study, a sample size estimation was performed for the COPD Assessment Test to detect a moderate effect size (f=0.30), with 80% power, 5% significance level and moderate correlation among repeated measures (r=0.25). The minimum sample size estimation was 36 participants. However, as in respiratory interventions dropout rates are around 30-35%, a total of 50 participants with AECOPD will be needed.

The plan is to recruit approximately 50 voluntary patients with AECOPD via clinicians at hospitals and primary care centres. This study will enroll adult patients diagnosed with AECOPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.

Patients will be recruited via the clinicians, who will provide a brief explanation about the study and inform the researcher about interested participants. Then, the researcher will contact interested participants and provide further information about the study, clarify any doubts and collect the inform consents. Patients will be eligible if they are: i) diagnosed with AECOPD according to the GOLD criteria; ii) included within 24-48h of the diagnostic; and iii) able to provide informed consent. Exclusion criteria will include: i) need for hospitalization; ii) other coexisting chronic respiratory diseases; iii) unstable cardiovascular disease; iv) musculoskeletal or neuromuscular conditions that preclude the performance of the assessments and/or treatment sessions; v) signs of cognitive impairment; vi) current neoplasia or immunological disease and vii) any therapeutic intervention in addition to standard of care.

Patients who agree to participate will be randomly allocated to the conventional treatment group (control group) or the conventional treatment plus PR group (experimental group).

Baseline data will be collected within the first 24-48 hours of the diagnosis of AECOPD. The researcher will collect sociodemographic, anthropometric and clinical data (e.g., number of exacerbations in the previous year); vital signs and peripheral oxygen saturation; symptoms (dyspnoea, fatigue, cough and sputum); lung function (spirometry); physical activity level; peripheral muscle strength (handgrip and hand-held dynamometer); functional status; exercise tolerance; impact of the disease and health-related quality of life.

Patients in the control group will receive daily medical treatment prescribed by the physician (i.e., medication).

Patients in the experimental group will receive daily medical treatment plus a community-based PR programme that will involve 6 sessions (2 times per week). The PR programme will consist of breathing retraining and airway clearance techniques, exercises for thoracic mobility, expansion and flexibility, cardiorespiratory exercise training, education and psychosocial support. This programme will be adjusted to each individual needs. After this period all measurements will be repeated. Furthermore, vital signs, peripheral oxygen saturation, dyspnoea and fatigue will also be collected before/during/after each session to monitor the intervention. Sessions will be conducted in properly equipped rooms or at patients' home and will last approximately 60 minutes.

Additionally, after 2, 6 and 12 months, the researcher will contact all participants via phone calls to collect data about the number of recurrent AECOPD, healthcare utilization (e.g., unscheduled visits, hospitalizations) and mortality.

Data analysis will be undertaken using Statistical Package for the Social Sciences (SPSS) software and will include descriptive and inferential statistics. To analyse changes in outcome measures, data from baseline and after treatment assessments will be compare. Moreover, between group comparisons will also be performed for baseline, after intervention and follow-ups assessments. Effect sizes for the interventions will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of AECOPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria (i.e., an episode of acute worsening of respiratory symptoms that result in additional therapy);
* included within 24-48h of the diagnostic;
* able to provide their own informed consent.

Exclusion Criteria:

* need for hospitalization;
* other coexisting chronic respiratory diseases;
* unstable cardiovascular disease;
* presence of musculoskeletal or neuromuscular conditions that preclude the performance of any of the assessments or the participation in the treatment sessions;
* signs of cognitive impairment;
* current neoplasia or immunological disease;
* any therapeutic intervention in addition to standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment test | 24-48 hours after hospital presentation or at clinical stabilization (baseline), after 3 weeks (after intervention) and after 2, 6 and 12 months at follow-ups.
  Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) is a short, simple, multidimensional, easy to administer and disease-specific questionnaire that measures impact of the disease. CAT consists of eight items (i.e., cough, sputum, chest tightness, breathlessness going up hills/stairs, activity limitations at home, confidence leaving home, sleep and energy) scored from 0 to 5. The individual score of each item is added to provide a total score that can range from 0 to 40. Total scores inferior to 10 are considered as "reduced impact", from 10-20 as "medium impact", from 21- 30 as "high impact" and above 30 as "very high impact". This is a valid and reliable instrument for use in patients with AECOPD (Chronbach's alpha=0.88).

SECONDARY OUTCOMES:
Physical activity level | assessment at baseline, after 3 weeks (after intervention) and after 2, 6 and 12 months at follow-ups
  Patients' physical activity level will be assessed with the brief physical activity assessment tool, which is a simple, quick and reliable instrument that is being validated for use in COPD and has been significantly correlated with the international physical activity questionnaire (r=0.523, p<0.001), accelerometers (r=0.529, p<0.001) and daily steps (r=0.565, p<0.001). It comprises two questions regarding the frequency and duration of moderate and vigorous physical activity undertaken in an usual week. Each question is scored from 0 to 4 and the total score consists of summing the result of the two questions, ranging from 0 to 8. Scores of 0-3 are considered "insufficiently active", and scores higher or equal to 4 "sufficiently active".
Symptoms of dyspnea | assessment at baseline and after 3 weeks (after intervention)
  Patients' self-reported level of dyspnea will be collected at rest, using the modified Borg scale. The level of dyspnea during activities will be collected with the modified British Medical Research Council questionnaire, which comprises five grades (statements) in a scale from 0 to 4, with higher grades indicating greater perceived respiratory limitation.
Symptoms of fatigue | assessment at baseline and after 3 weeks (after intervention)
  Patients' self-reported level of fatigue will be collected at rest, using the modified Borg scale. The level of fatigue on a daily basis will be collected with the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) and the Checklist of Individual Strength 8 (CIS-8).
Lung function measurement | assessment at baseline and after 3 weeks (after intervention)
  A spirometry test will be performed with a portable spirometer to assess the force expiratory volume in 1 second and, therefore, the degree of bronchial obstruction.
Change in muscle strength | assessment at baseline and after 3 weeks (after intervention)
  Patients' handgrip, biceps and quadriceps muscle strength will be collected with a hand-held dynamometer.
Change in functional status | assessment at baseline and after 3 weeks (after intervention)
  Patients' functional level will be assessed with the short physical performance battery, a simple and easy to perform tool that includes the four-meter gait speed test, the five-repetition sit-to-stand test and a balance test, and gives a total score based on the performance in each of those tests.
1-minute sit-to-stand test | assessment at baseline and after 3 weeks (after intervention)
  The 1-minute sit-to-stand test will be used to also assess functional status.
Change in exercise capacity | assessment at baseline and after 3 weeks (after intervention)
  Patients' exercise capacity will be assessed using the Chester step test, since it allows exercise prescription and is feasible in the community and at patients' home. Additionally, patients assessed in the community, at the facilities of University of Aveiro, will also perform the 6-minutes walk test to assess their exercise capacity.
London Chest Activities of Daily Living | assessment at baseline and after 3 weeks (after intervention)
  Patients' level of dyspnoea performing activities of daily living and functional status will be assessed with th London Chest Activities of Daily Living questionnaire.
Cough And Sputum Assessment Questionnaire | assessment at baseline and after 3 weeks (after intervention)
  Patients' symptoms of cough and sputum will be assessed with the Cough And Sputum Assessment Questionnaire (CASA-Q).
Number of hospitalizations | assessment at baseline and after 2, 6 and 12 months from the end of the intervention (follow-ups)
  Patients' number of hospitalizations in the previous year and during the follow-up period after the acute exacerbation will be assessed by asking the patient to self-report it.
Re-exacerbations | assessment at baseline and after 2, 6 and 12 months from the end of the intervention (follow-ups)
  Patients' number of re-exacerbations after being included in the study will be assessed by asking the patient to self-report it.
Mortality | assessment at baseline and after 2, 6 and 12 months from the end of the intervention (follow-ups)
  The number of patients who died after the acute exacerbation, up to the 1 year follow-up period, will be collected.

OTHER OUTCOMES:
Body mass index | assessment at baseline
  Patients' body mass index will be assessed in kg/m^2 based on patients' height and weight.
Heart rate | assessment at baseline and 3 weeks after intervention
  Heart rate will be assessed in beats per minute using a oximeter and blood pressure meter.
Respiratory rate | assessment at baseline and 3 weeks after intervention
  Respiratory rate will be assessed by direct observation, counting the number of respiratory cycles.
Blood pressure | assessment at baseline and 3 weeks after intervention
  Blood pressure will be assessed using a blood pressure meter.
Peripheral Oxygen Saturation | assessment at baseline and 3 weeks after intervention
  Peripheral oxygen saturation will be assessed with a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira A, Machado A, Marques A. Minimal Important and Detectable Differences of Respiratory Measures in Outpatients with AECOPDdagger. COPD. 2018 Oct;15(5):479-488. doi: 10.1080/15412555.2018.1537366. Epub 2018 Dec 4. PMID 30512981
- [Background] Oliveira A, Marques A. Understanding symptoms variability in outpatients with AECOPD. Pulmonology. 2018 Nov-Dec;24(6):357-360. doi: 10.1016/j.pulmoe.2018.09.007. No abstract available. PMID 30554671
- [Background] Oliveira A, Afreixo V, Marques A. Enhancing our understanding of the time course of acute exacerbations of COPD managed on an outpatient basis. Int J Chron Obstruct Pulmon Dis. 2018 Nov 20;13:3759-3766. doi: 10.2147/COPD.S175890. eCollection 2018. PMID 30538438
- [Background] Oliveira AL, Marques AS. Outcome Measures Used in Pulmonary Rehabilitation in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Systematic Review. Phys Ther. 2018 Mar 1;98(3):191-204. doi: 10.1093/ptj/pzx122. PMID 29228288
- [Background] Oliveira A, Marques A. Exploratory mixed methods study of respiratory physiotherapy for patients with lower respiratory tract infections. Physiotherapy. 2016 Mar;102(1):111-8. doi: 10.1016/j.physio.2015.03.3723. Epub 2015 May 14. PMID 26067286
- [Background] Oliveira A, Pinho C, Marques A. Effects of a respiratory physiotherapy session in patients with LRTI: a pre/post-test study. Clin Respir J. 2017 Nov;11(6):703-712. doi: 10.1111/crj.12402. Epub 2015 Nov 5. PMID 26471240
- [Background] Machado A, Oliveira A, Valente C, Burtin C, Marques A (2018) "Community-based pulmonary rehabilitation during acute exacerbations of COPD" European Respiratory Journal
- [Background] Machado A, Silva P, Marques A (2018) "Design of pulmonary rehabilitation during acute exacerbations of COPD". European Respiratory Journal
- [Background] Oliveira A, Rebelo P, Andrade L, Valente C, Marques A (2018) "Computerised respiratory sounds during acute exacerbations of Chronic Obstructive Pulmonary Disease". Proceedings of the 4th IPLeiria's International Health Congress. BMC Health Services Research 2018, 18(Suppl 2): O23 pp 13
- [Background] Machado A, Oliveira A, Paixão C, Miranda S, Melro H, Ferreira D, Marques A (2017) "Pulmonary rehabilitation effects on computerized respiratory sounds of patients with AECOPD" Proceedings of the 42nd Annual Conference of the International Lung Sound Association, 182:57
- [Background] Machado A, Oliveira A, Valente C, Burtin C, Marques A. Effects of a community-based pulmonary rehabilitation programme during acute exacerbations of chronic obstructive pulmonary disease - A quasi-experimental pilot study. Pulmonology. 2020 Jan-Feb;26(1):27-38. doi: 10.1016/j.pulmoe.2019.05.004. Epub 2019 Jun 1. PMID 31164288
- [Background] Machado A, Oliveira A, Valente C, Burtin C, Marques A. Effects of a community-based pulmonary rehabilitation programme during acute exacerbations of chronic obstructive pulmonary disease - A quasi-experimental pilot study. Authors' reply. Pulmonology. 2020 Mar-Apr;26(2):112-113. doi: 10.1016/j.pulmoe.2019.09.001. Epub 2019 Oct 8. No abstract available. PMID 31601490
- [Derived] Machado A, Dias C, Paixao C, Goncalves AP, Burtin C, Marques A. Short-term effects of home-based pulmonary rehabilitation during outpatient-managed exacerbations of COPD: a randomised controlled trial. Thorax. 2025 Mar 18;80(4):218-226. doi: 10.1136/thorax-2024-221760. PMID 39689939